CLINICAL TRIAL: NCT00535899
Title: Speckle Tracking Imaging in Patients With Low Ejection Fraction Aortic Stenosis (SPArKLE-AS)
Acronym: SPArKLE-AS
Status: Terminated | Type: Observational
Why Stopped: unable to find subjects meeting inclusion criteria
Sponsor: The Cleveland Clinic (Other)
Other Study IDs: 07-578
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Last update posted 2008-05-26 (Estimated); Status verified 2008-05

CONDITIONS: Aortic Stenosis
Keywords: Aortic stenosis; Speckle tracking imaging; Low ejection fraction; Aortic valve replacement; Strain
MeSH Terms: conditions — Aortic Valve Stenosis; Sprains and Strains

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In patients with aortic stenosis and low ejection fraction, how can we predict who will recover their ejection fraction after aortic valve replacement? We plan to observe 50 patients with Low EF aortic stenosis and perform serial echocardiograms pre and post-aortic valve replacement and analyze regional wall motion contractility with a new software application called speckle tracking imaging.

DETAILED DESCRIPTION:
In patients with severe aortic stenosis and LV dysfunction, 76% of patients have an improvement of ventricular function and NYHA class, after aortic valve replacement. The prognostic indicators of which patients will recover EF post-operatively, has not been fully established, but has been linked to a history of prior MI and pre-operative aortic valve area. Furthermore it is hypothesized that those ventricles that do not recover are fibrosed, either from prior MI or long standing LVH (hypertrophy).

Currently systolic and diastolic function will be measured pre-operatively with standard 2D echo and Doppler. 2D Strain and Strain rate imaging with speckle tracking is a novel method of assessing regional as well as global "contractility". This method overcomes many limitations inherent in assessing myocardial functioning with current methodology, mainly it is reproducible, objective, and is independent of myocardial translation, tethering and furthermore as speckle tracking is derived from B mode images is independent of Doppler angle.The applicability of this technology to patients with aortic valve stenosis and systolic dysfunction and its clinical significance has not been evaluated. We hypothesize that patients with reduced peak systolic strain rate and diastolic strain rates at baseline adjusted for LVEF will have poorer recovery of LVEF than those with relatively preserved strain or strain rate. As this is a pilot study, we plan to prospectively analyze 50 consecutive patients who have severe aortic stenosis and left ventricular systolic dysfunction, EF under 40% with Speckle imaging derived strain rate imaging pre and post-operatively for aortic valve replacement. This would be done as part of routine pre-operative and post-operative transthoracic echocardiography using standard views, with the exception that all studies would need to be done on the GE Vivid 7 digital ultrasound system. Speckle derived imaging data is derived from standard B mode (Grey scale images), with a frame rate of 50 f/s. 3 D images will also be obtained. Post-operative TTE's will be performed before discharge and 4-12 months+/- 30 days after discharge. Baseline characteristics will be taken from the standard pre-operative baseline study including basic 2 D valve area, EF, wall thickness and geometry, and Doppler flow data. Exclusion criteria: Patients with prior cardiac surgery including CABG or other valve replacement, more than mild mitral valve or aortic regurgitation and chronic kidney disease (Cr 1.5), emergent aortic valve replacement, or endocarditis, or CAD on LHC > 50%. Informed consent will be obtain on all patients, and they will only be included if they consent. No surgery will be delayed for purpose of the study if the proper hardware/GE VIVID system is not available.

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic stenosis with ejection fraction less than 40% that is schedule to undergo aortic valve replacement

Exclusion Criteria:

* Creatinine > 2
* More than moderate mitral, tricuspid, or aortic regurgitation.
* Endocarditis
* Emergent surgery
* Prior sternotimy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-09

CONTACTS AND LOCATIONS:
Overall Officials: Ryan P Daly, MD, Principal Investigator — CCF
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States